CLINICAL TRIAL: NCT00614536
Title: Observational Study: Changes in Reflux Symptoms and Reflux Finding Score According to Rabeprazole Treatment Period
Brief Title: Study of Changes in Reflux Symptoms and Reflux Finding Score According to Rabeprazole Treatment Period
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR014812
Record Dates: First submitted 2008-01-24; First posted 2008-02-13 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Gastroesophageal Reflux; Pharyngeal Diseases
Keywords: Reflux Symptom Index; Reflux Finding Score; Rabeprazole; LaryngoPharyngeal Reflux Disease; GastroEsophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux; Pharyngeal Diseases | interventions — Rabeprazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001
  Interventions: Drug: Rabeprazole Sodium

INTERVENTIONS:
Drug: Rabeprazole Sodium — 10mg - 20mg tablet once or twice daily for 12weeks

SUMMARY:
The purpose of this observational study is to examine RSI (Reflux Symptom Index) and RFS (Reflux Finding Score) by treatment period before and after rabeprazole treatment in LaryngoPharyngeal Reflux Disease(LPRD) patients.

DETAILED DESCRIPTION:
This clinical study is a multicenter, open-label, prospective, observational study of outpatients who visit the department of otolaryngology (branch of medicine that deals with diagnosis and treatment of diseases of the ear, nose, and throat) under routine practice. This study will examine RSI (Reflux Symptom Index) and RFS (Reflux Finding Score) by treatment period (before and after rabeprazole treatment) in patients with LaryngoPharyngeal Reflux Disease(LPRD). Among the patients who visit the department of otolaryngology with suspicious laryngopharyngeal reflux, those needing rabeprazole sodium treatment according to the doctor's discretion are eligible for enrollment. This study will explore the correlation between RSI and RFS and will examine major reflux symptoms and types of lesions, to find the most reliable factors in diagnosing LPRD and judging therapeutic effectiveness of treatments. LPRD is a disease with various symptoms and causes lesions by exposing the upper respiratory system to gastric acid and stomach contents. RSI and RFS can be used to diagnose LPRD in a relatively objective manner by scoring items of symptoms and lesions particular to LPRD. Evaluations will be performed four times from baseline to week 12. Observational Study - one tablet of rabeprazole 10 mg or 20 mg once daily for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients who visit the department of otolaryngology with suspicious laryngopharyngeal reflux
* Patients who need rabeprazole treatment according to the doctor's discretion
* Patients who have signed an informed consent document indicating that they understand the purpose of and procedures required for the observational study and they agree to provide their information

Exclusion Criteria:

* Patients who took rabeprazole within the past one month
* Patients who are hypersensitive to any of rabeprazole or benzimidazole
* Patients with severe hepatic impairment
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among the patients who visit the department of otolaryngology with suspicious laryngopharyngeal reflux ; Patients who need rabeprazole treatment according to the doctor's discretion
Sampling Method: Non-Probability Sample
Enrollment: 1142 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The change from baseline in RSI and RFS score during LPRD treatment period, | 12 weeks

SECONDARY OUTCOMES:
Regional difference in distribution of symptoms and lesions, and in severity | 12 weeks
LRPD treatment period with rabaprazole sodium | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.